CLINICAL TRIAL: NCT04094194
Title: Relation of the Nordic Dietary Pattern With Cardiometabolic Risk Factors and Incident Cardiovascular Outcomes: A Systematic Review and Meta-analysis of Randomized Controlled Trials and Prospective Cohort Studies
Brief Title: Meta-analysis of the Nordic Dietary Pattern on Cardiometabolic Risk and Cardiovascular Outcomes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canada Research Chairs Endowment of the Federal Government of Canada (Other Government); The Physicians' Services Incorporated Foundation (Other); Canadian Diabetes Association (Other)
Responsible Party: Principal Investigator, John Sievenpiper, MD, PhD, FRCPC, University of Toronto
Other Study IDs: DNSG-Nordic diet
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Body Weight; Obesity; Overweight and Obesity; Obesity, Abdominal; Hypertension; Hyperlipidemias; Cardiovascular Diseases; Coronary Heart Disease; Stroke; Mortality; Dyslipidemias; Diabetes; PreDiabetes; Insulin Tolerance; Dysglycemia; Metabolic Syndrome
Keywords: Nordic diet; Cardiometabolic risk factors; Mortality; Cardiovascular diseases; Type 2 diabetes; Hypertension; Systematic review and meta-analysis; Randomized controlled trials; Prospective cohort studies
MeSH Terms: conditions — Body Weight; Obesity; Overweight; Obesity, Abdominal; Hypertension; Hyperlipidemias; Cardiovascular Diseases; Coronary Disease; Stroke; Dyslipidemias; Diabetes Mellitus; Prediabetic State; Metabolic Syndrome; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nordic diet — Healthy dietary pattern that is consumed in Nordic countries

SUMMARY:
The Nordic Diet is a dietary pattern rich in traditional Nordic foods, including berries, grains, and fatty fish common in northern Europe. Studies have shown a protective effect of the Nordic Diet on cardiometabolic risk factors, however only select clinical practice guidelines for the management of diabetes (i.e. Diabetes Canada) recommend this dietary pattern. To support the update of the EASD clinical practice guidelines for nutrition therapy, the investigators propose to conduct a systematic review and meta-analysis of prospective cohort studies and clinical trials to investigate the association between the Nordic Diet, cardiometabolic outcomes and cardiovascular disease incidence and mortality. The findings generated by this proposed knowledge synthesis will help improve the health of consumers through informing evidence-based guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

DETAILED DESCRIPTION:
Background: Greater adherence to the Mediterranean diet, a traditional dietary pattern of the wider region of the Mediterranean sea, has been associated with favourable cardiometabolic outcomes, including the prevention of type 2 diabetes and cardiovascular diseases (CVD). However, limited local food availability, increased cost or unfamiliar culture and tradition render the Mediterranean diet difficult to follow in the northern European environment. The Nordic Diet or those of other traditional diets of the Nordic countries (Sweden, Norway, Finland, Denmark, Iceland, Faeroe islands) are dietary patterns rich in traditional Nordic foods, including berries, grains, and fatty fish common in northern Europe. The Nordic Diet has been associated with favorable cardiometabolic outcomes including improved lipid profile and insulin sensitivity. These benefits have been recognized in the most recent updates of the clinical practice guidelines for diabetes in Canada. The European Association for the Study of Diabetes (EASD) has not included the Nordic dietary pattern in their guidelines.

Need for proposed research: High quality systematic reviews and meta-analyses of randomized controlled trials and prospective cohorts represent high-quality evidence to support dietary guidelines and public health policy. As dietary guidelines and public health policy have shifted towards food and dietary-pattern based recommendations, there is a need for systematic reviews and meta-analyses comparing the role of the Nordic diet in the prevention and management of cardiometabolic outcomes and cardiovascular diseases.

Objectives: To support the update of the European Association for the Study of Diabetes (EASD) clinical practice guidelines for nutrition therapy, the investigators will conduct a systematic review and meta-analysis of randomized controlled trials and prospective cohorts using the GRADE approach on the Nordic dietary pattern on cardiometabolic risk factors and cardiovascular disease outcomes.

Design: The systematic review and meta-analysis of clinical trials and prospective cohort studies will be conducted according to the Cochrane Handbook for Systematic Reviews of interventions and reported according to the Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA) and Meta-analysis of Observational Studies in Epidemiology (MOOSE) guidelines.

Data sources: MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms supplemented by hand searches of references of included studies.

Study selection: Randomized controlled trials conducted in humans with a follow-duration ≥ 3 week investigating the effect of a Nordic diet on cardiometabolic outcomes will be included. Studies that are not conducted in humans, not randomized, have an acute feeding design (<3 weeks), lack a suitable control (non-isocaloric) and/or do not report viable endpoint data will not be included. Prospective cohort studies with greater than 1-year of follow-up will be included.

Data extraction: Two or more investigators will independently extract relevant data and assess risk of bias using the Cochrane Risk of Bias Tool for randomized clinical trials and the Newcastle Ottawa Scale for prospective cohorts. All disagreements will be resolved by consensus. Standard computations and imputations will be used to derive missing variance data for the randomized clinical. Risk ratios, odds ratios and hazard ratios for clinical outcomes in the prospective cohort studies will be extracted or derived from clinical event data across exposure to a Nordic diet.

Outcomes: For the randomized clinical trials, the primary outcome will be LDL-cholesterol. Secondary outcomes will include markers of glycemic control (HbA1c, fasting glucose, fasting insulin); other blood lipids (non-HDL-C, apo B, HDL-C, triglycerides); adiposity (body weight, BMI, waist circumference), blood pressure (systolic and diastolic blood pressure) and inflammation (C-reactive protein [CRP]).

For prospective cohorts, the primary outcome will be incident CVD Secondary outcomes include incident coronary heart disease (CHD) and incident stroke.

Data synthesis:

Trials: Data will be pooled by the generic inverse-variance method with DerSimonian and Laird random-effects models and expressed as mean differences (MDs) with 95% confidence intervals (95% CIs). Random-effects models were used as they account for residual heterogeneity and yield more conservative estimates. Fixed-effects models will be used for <5 trials. Paired analyses will be applied to all crossover trials. Heterogeneity will be tested by Cochran's Q statistic and quantified by the I2 statistic. To explore sources of heterogeneity, we will conduct sensitivity analyses, in which each study is systematically removed. If there are ≥10 trials, we will explore sources of heterogeneity by a priori subgroup analyses by study design (parallel or crossover), follow-up duration (<12 weeks or ≥12 weeks), comparator diet, baseline measurements, risk of bias, disease duration, and funding source. Significant unexplained heterogeneity will be investigated by additional post hoc subgroup analyses (e.g. age, sex, diet quality index, composition of the background diet [total % energy from fat, carbohydrate, protein]). Meta-regression analyses will assess the significance of categorical and continuous subgroups analyses. When ≥10 studies are available, publication bias will be investigated by inspection of funnel plots and formal testing using the Egger and Begg tests. If publication bias is suspected, we will attempt to adjust for funnel plot asymmetry by imputing the missing study data using the Duval and Tweedie trim and fill method.

Prospective cohort studies: Natural log-transformed relative risks (RRs) or hazard ratios (HRs) of clinical outcomes, comparing extreme quantiles (the highest exposure versus the lowest exposure or reference group), will be pooled separately using the generic inverse variance method with random effects models and expressed as RRs with 95% confidence intervals (CIs). Heterogeneity will be tested by Cochran's Q statistic and quantified by the I2 statistic. To explore sources of heterogeneity, we will conduct sensitivity analyses, in which each study is systematically removed. If ≥10 cohort comparisons were available, then we will perform an a-priori subgroup analyses by meta-regression for follow-up (<10 years vs. ≥10 years), sex (males vs. females, males vs. mixed, females vs. mixed), study quality (NOS <6 vs. ≥6) and funding source. Significant unexplained heterogeneity will be investigated by additional post hoc subgroup analyses. Linear and non-linear dose-response relations will be explored with the use of random-effects generalised least-squares trend estimation (GLST) models and spline curve modeling (MKSPLINE procedure), respectively. When ≥10 studies are available, publication bias will be investigated by inspection of funnel plots and formal testing using the Egger and Begg tests. If publication bias is suspected, we will attempt to adjust for funnel plot asymmetry by imputing the missing study data using the Duval and Tweedie trim and fill method.

Evidence assessment: The certainty of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE).

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition, diabetes, obesity, and cardiovascular disease. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Significance: The proposed project will aid in knowledge translation to the role of the Nordic Diet in cardiovascular disease prevention and management, strengthening the evidence-base for guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria for controlled trials:

* dietary trials in humans
* Nordic diets intervention
* Presence of an adequate comparator (ad libitum control)
* Diet duration >=3 weeks
* Viable outcome data

Inclusion Criteria for prospective cohort studies:

* Prospective cohort studies
* Duration >= 1 year
* Assessment of the exposure of a Nordic Diet
* Ascertainment of viable data by level of exposure

Exclusion Criteria for controlled trials:

* Non-human trials
* Observational studies
* Lack of suitable comparator diet (i.e. non-isocaloric)
* Diet duration <3-weeks
* No viable outcome data

Exclusion Criteria for prospective cohort studies:

* Ecological, cross-sectional, retrospective observational studies, clinical trials, and non-human studies
* Duration < 1 year
* non assessment of exposure of a Nordic diet
* No ascertainment viable clinical outcome data by level of exposure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals, both children, and adults, regardless of health status.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Incident Cardiovascular Disease (Prospective Cohort Studies) | Time Frame: At least 1 year
  Relative Risks
LDL-cholesterol (randomized and non-randomized controlled trials) | Time Frame: Up to 20 years
  Mean difference

SECONDARY OUTCOMES:
Glycemic control - Fasting blood glucose (randomized and non-randomized controlled trials) | Time Frame: Up to 20 years
  Mean Difference
Glycemic control - HbA1c (randomized and non-randomized controlled trials) | Time Frame: Up to 20-years
  Mean Difference
Glycemic control - Fasting insulin (randomized and non-randomized controlled trials) | Time Frame: Up to 20-years
  Mean Difference
Blood lipids - non-HDL-cholesterol (randomized and non-randomized controlled trials) | Time Frame: Up to 20-years
  Mean Difference
Blood lipids - HDL-cholesterol (randomized and non-randomized controlled trials) | Time Frame: Up to 20-years
  Mean difference
Blood lipids - Triglycerides (randomized and non-randomized controlled trials) | Time Frame: Up to 20-years
  Mean Difference
Blood lipids - apo B (randomized and non-randomized controlled trials) | Time Frame: Up to 20-years
  Mean Difference
Adiposity - Body mass index (BMI) (randomized and non-randomized controlled trials) | Time Frame: Up to 20-years
  Mean Difference
Adiposity - Body weight (randomized and non-randomized controlled trials) | Time Frame: Up to 20-years
  Mean Difference
Adiposity - Waist circumference (randomized and non-randomized controlled trials) | Time Frame: Up to 20-years
  Mean Difference
Blood pressure - systolic blood pressure (randomized and non-randomized controlled trials) | Time Frame: Up to 20-years
  Mean Difference
Blood pressure - diastolic blood pressure (randomized and non-randomized controlled trials) | Time Frame: Up to 20-years
  Mean Difference
Inflammation - C-reactive protein (CRP) (randomized and non-randomized controlled trials) | Time Frame: Up to 20-years
  Mean Difference
Incident Coronary Heart Disease (Prospective Cohort Studies) | Time Frame: At least 1 year
  Relative Risks
Incident Stroke (Prospective Cohort Studies) | Time Frame: At least 1 year
  Relative Risks

CONTACTS AND LOCATIONS:
Overall Officials: John Sievenpiper, MD,PhD,FRCPC, Principal Investigator — University of Toronto
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Salas-Salvado J, Bullo M, Babio N, Martinez-Gonzalez MA, Ibarrola-Jurado N, Basora J, Estruch R, Covas MI, Corella D, Aros F, Ruiz-Gutierrez V, Ros E; PREDIMED Study Investigators. Reduction in the incidence of type 2 diabetes with the Mediterranean diet: results of the PREDIMED-Reus nutrition intervention randomized trial. Diabetes Care. 2011 Jan;34(1):14-9. doi: 10.2337/dc10-1288. Epub 2010 Oct 7. PMID 20929998
- [Background] Fung TT, Rexrode KM, Mantzoros CS, Manson JE, Willett WC, Hu FB. Mediterranean diet and incidence of and mortality from coronary heart disease and stroke in women. Circulation. 2009 Mar 3;119(8):1093-100. doi: 10.1161/CIRCULATIONAHA.108.816736. Epub 2009 Feb 16. PMID 19221219
- [Background] Papadaki A, Scott JA. The impact on eating habits of temporary translocation from a Mediterranean to a Northern European environment. Eur J Clin Nutr. 2002 May;56(5):455-61. doi: 10.1038/sj.ejcn.1601337. PMID 12001018
- [Background] Adamsson V, Reumark A, Cederholm T, Vessby B, Riserus U, Johansson G. What is a healthy Nordic diet? Foods and nutrients in the NORDIET study. Food Nutr Res. 2012;56. doi: 10.3402/fnr.v56i0.18189. Epub 2012 Jun 27. PMID 22761599
- [Background] Adamsson V, Reumark A, Fredriksson IB, Hammarstrom E, Vessby B, Johansson G, Riserus U. Effects of a healthy Nordic diet on cardiovascular risk factors in hypercholesterolaemic subjects: a randomized controlled trial (NORDIET). J Intern Med. 2011 Feb;269(2):150-9. doi: 10.1111/j.1365-2796.2010.02290.x. Epub 2010 Oct 22. PMID 20964740
- [Background] Roswall N, Sandin S, Scragg R, Lof M, Skeie G, Olsen A, Adami HO, Weiderpass E. No association between adherence to the healthy Nordic food index and cardiovascular disease amongst Swedish women: a cohort study. J Intern Med. 2015 Nov;278(5):531-41. doi: 10.1111/joim.12378. Epub 2015 May 19. PMID 25991078
- [Background] Kanerva N, Kaartinen NE, Rissanen H, Knekt P, Eriksson JG, Saaksjarvi K, Sundvall J, Mannisto S. Associations of the Baltic Sea diet with cardiometabolic risk factors--a meta-analysis of three Finnish studies. Br J Nutr. 2014 Aug 28;112(4):616-26. doi: 10.1017/S0007114514001159. Epub 2014 May 27. PMID 24867656
- [Derived] Massara P, Zurbau A, Glenn AJ, Chiavaroli L, Khan TA, Viguiliouk E, Mejia SB, Comelli EM, Chen V, Schwab U, Riserus U, Uusitupa M, Aas AM, Hermansen K, Thorsdottir I, Rahelic D, Kahleova H, Salas-Salvado J, Kendall CWC, Sievenpiper JL. Nordic dietary patterns and cardiometabolic outcomes: a systematic review and meta-analysis of prospective cohort studies and randomised controlled trials. Diabetologia. 2022 Dec;65(12):2011-2031. doi: 10.1007/s00125-022-05760-z. Epub 2022 Aug 26. PMID 36008559